CLINICAL TRIAL: NCT02491736
Title: Ketoprofen Gel vs Placebo in Children Presented With Ankle Sprain to the Emergency Department: A Randomised Controlled Trial
Brief Title: Ketoprofen Gel vs Placebo in Children With Ankle Sprain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16445
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketoprofen (Experimental): 2.5% ketoprofen gel
  Interventions: Drug: Ketoprofen
- Placebo (Placebo Comparator): Placebo gel
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ketoprofen — 2.5% ketoprofen gel
  Other Names: Fastjel
  Arms: ketoprofen
Other: Placebo — Placebo gel
  Arms: Placebo

SUMMARY:
The aim of this study is to analyse the effect of ketoprofen gel in children presented with ankle sprain to the emergency department.

DETAILED DESCRIPTION:
Ankle sprains may be associated with soft tissue injuries and fractures. Although diagnostic modalities are important, alleviation of pain is also a part of emergency department management. The aim of this study is to analyse the effect of ketoprofen gel in children presented with ankle sprain to the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ankle sprain
* Patients over 8 and lower than 18 years old

Exclusion Criteria:

* Ankle sprain more than 24 hours
* visual analogue scale score lower than 40mm
* Allergy to the study drug

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 30 minutes
  Measurement of pain reduce at 30 minutes by visual analogue scale

SECONDARY OUTCOMES:
Adverse effects | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Serinken, MD, Study Chair — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)